CLINICAL TRIAL: NCT06287333
Title: Video-respiratory Polygraphy for the Diagnosis of Obstructive Sleep Apnea Syndrome in Children
Brief Title: Video-respiratory Polygraphy in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI221
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: child; polysomnography; polygraphy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography in routine care — Children performed a polysomnography in routine clinical care

SUMMARY:
The diagnosis of obstructive sleep apnea-hypopnea syndrome in children (OSAS) requires a polysomnography (PSG) in a sleep lab with video surveillance and monitoring by a nurse. But PSG is a cumbersome exam, sometimes difficult to perform in children. Simplified exams as respiratory polygraphy (RP) which uses only respiratory signals can be used for the diagnosis of OSAS but studies show that it underestimates the obstructive apnea-hypopnea index (OAHI) because the total sleep time cannot be accurately estimated. The use of a video camera with software synchronous with the RP software could compensate for this disadvantage, by estimating when the child is sleeping or not.

DETAILED DESCRIPTION:
The diagnosis of obstructive sleep apnea-hypopnea syndrome in children (OSAS) requires the performance of a polysomnography (PSG) in a sleep lab with video surveillance and monitoring by a nurse to put the sensors back on the child if necessary. PSG gives the obstructive apnea-hypopnea index (OAHI) necessary for the diagnosis of OSA and to determine its severity. But PSG is a cumbersome exam, sometimes difficult to carry out in children, with several sensors and electrodes to install (electroencephalogram (EEG), myogram (EMG), occulogram (EOG), necessary to determine awakening and sleep periods and intra-sleep micro-arousals, nasal cannula, thoraco-abdominal straps, pulse oximetry, actimetry to score respiratory events). PSG is time-consuming for installation and analysis. Simplified methods of recording and analysis are preferable in children but require validation in this population.

Respiratory polygraphy (RP) which uses only respiratory signals (without EEG, EMG and EOG) can be used for the diagnosis of OSA but studies showed that it underestimated the OAHI because the total sleep time cannot be accurately estimated. The use of a video camera with software synchronous with the RP software could compensate for this disadvantage, by estimating when the child is sleeping or not.

The hypothesis of this study is that video-RP can identify OSAS in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with suspicion of OSAS
* Interpretable polysomnography

Exclusion Criteria:

* Non-interpretable polysomnography

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 2 to 19 years adressed for a PSG in routine clinical care for suspicion of OSAS by the ear-nose-throat physician, pediatric pulmonologist, sleep specialist, endocrinologist, genetician.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
OAHI in video-RP significantly correlated with OAHI in PSG | One night
  Value of the OAHI obtained by the video-RP for each of the children in the groups with OSAS (who have an OAHI ≥ 1/h in PSG) and without OSAS (who have an OAHI < 1/h in PSG) will be correlated with the value of OAHI obtained by PSG using a Fisher exact test

SECONDARY OUTCOMES:
Diagnostic ability of video-RP to identify OSAS in children | One night
  ROC curves to determine the sensitivity and specificity of the OAHI obtained by video-RP to identify children with OSA
Diagnostic ability of video-RP to identify moderate-severe OSAS in children | One night
  ROC curves to determine the sensitivity and specificity of the OAHI obtained by video-RP to identify children with moderate-severe OSA (with an OAHI ≥ 5 /h in PSG)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Horne AF, Olafsdottir KA, Arnardottir ES. In-person vs video hookup instructions: a comparison of home sleep apnea testing quality. J Clin Sleep Med. 2022 Aug 1;18(8):2069-2074. doi: 10.5664/jcsm.10084. PMID 35510598
- [Result] Sivan Y, Kornecki A, Schonfeld T. Screening obstructive sleep apnoea syndrome by home videotape recording in children. Eur Respir J. 1996 Oct;9(10):2127-31. doi: 10.1183/09031936.96.09102127. PMID 8902478